CLINICAL TRIAL: NCT04460183
Title: An Open-label, Adaptive Randomized, Controlled Multicenter Study to Evaluate the Efficacy and Safety of RESP301 Plus Standard of Care (SOC) Compared to SOC Alone in Hospitalized Participants With COVID-19 WHO Grade 3&4 (NOCoV2)
Brief Title: A Study to Assess Efficacy and Safety of RESP301 Plus Standard of Care (SOC) Compared to SOC Alone in Hospitalized Participants With COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Thirty Respiratory Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESP301-002
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational arm (Experimental): Participants will receive inhaled RESP301 administered using a nebulizer three times a day for up to 10 days in addition to the standard of care.
  Interventions: Drug: RESP301, a Nitric Oxide generating solution; Other: Standard of Care
- Control arm (Active Comparator): Participants will receive institutional SOC for the treatment of COVID-19
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: RESP301, a Nitric Oxide generating solution — Product application requires inhalation using a standard handheld nebulizer.
  Arms: Investigational arm
Other: Standard of Care — Participants will receive institutional SOC for the treatment of COVID-19.

SUMMARY:
The effect of RESP301 as an add on treatment to SOC will be evaluated for its efficacy in reducing rate of progression to a more severe level of COVID-19 and for safety, by comparison with SOC alone in hospitalized COVID-19 patients.

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter, parallel group, concurrent, controlled study using a sequential adaptive design to evaluate the efficacy and safety of RESP301 plus SOC versus SOC alone in hospitalized patients with COVID-19 (World Health Organization [WHO] ordinal scale level 3 or 4).

Approximately 300 participants will be enrolled and randomized 2:1 to the Investigational arm or the Control arm. The study will be divided into the following periods: Screening period: (up to 2 days), Intervention (up to 10 days), follow-up (Day 14 and Day 28).

ELIGIBILITY:
Inclusion Criteria:

1. Participant has laboratory-confirmed SARS-CoV-2 infection as determined by reverse transcriptase polymerase chain reaction (RT-PCR) or other approved clinical testing prior to randomization.
2. Participant is hospitalized in relation to COVID-19, requiring supplemental oxygen to maintain SpO2 at a safe level (WHO level 3 & 4).
3. Participant is capable of giving signed informed consent
4. Participant is male or female. All females of childbearing potential, including pregnant females, must consent to urine pregnancy testing at screening to be eligible for the study.

Exclusion Criteria:

1. Rapidly deteriorating or likely to require escalation to high flow oxygen, invasive or non-invasive ventilatory support within 24 hours according to Investigator's opinion.
2. Unable to safely receive a nebulized treatment for approximately 8 minutes according to Investigator's opinion.
3. Unable to receive or considered ineligible for invasive or non-invasive ventilatory support.
4. History of methemoglobinemia.
5. Presence of uncontrolled asthma, history of severe bronchospasm.
6. Presence of severe chronic respiratory disease and tracheostomy.
7. Suspected or confirmed untreated, active tuberculosis.
8. Severely immune-compromised participants in Investigator's opinion.
9. Recent active coronary artery disease or decompensated heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, St. Mary's Hospital, London
  - Royal Preston Hospital, Preston

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 centers that enrolled 19 participants in the United Kingdom (UK) from 29-Jul-2020 (First Enrolment) to 21-May-2021 (Last Participant Completed).
Pre-assignment Details: The screening period was of 2 days. All the study assessments were performed as per the schedule of assessment.
Groups:
- RESP301+SoC: Participants received inhaled RESP301 administered using a nebulizer three times a day (TID) for up to 10 days in addition to the standard of care (SoC).
- Standard of Care (SoC): Participants received institutional SOC alone for the treatment of COVID-19.
Period: Overall Study
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Started | 14 | 5
Completed | 10 | 4
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RESP301+SoC | Standard of Care (SoC) | Total
Number analyzed (Participants) | 14 | 5 | 19
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 11 | 4 | 15
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 4 | 18
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Progress by at Least One Level Higher on the Modified WHO Ordinal Scale
Description: A modified WHO ordinal scale was used for consistency with the recent study in adults hospitalized with severe COVID-19, to record the participant's status at the time of assessment. The modified WHO ordinal scale included the following levels :
  1= Not hospitalized, no limitations on activities; 2= Not hospitalized, limitation on activities; 3= Hospitalized, not requiring supplemental oxygen; 4= Hospitalized, requiring supplemental oxygen; 5= Hospitalized, on non-invasive ventilation or high-flow oxygen devices; 6= Hospitalized, on invasive mechanical ventilation or extra corporeal membrane oxygenation (ECMO); 7= Death. Higher scores mean worse outcome. The number of participants that had an increase in at least one level higher score on the modified WHO ordinal scale was assessed.
Time Frame: Baseline, Day 2 and Day 3
Population: The intent-to-treat (ITT) population included all randomized participants. For RESP301+SoC arm only 1 participant was available for this analysis who had an increase in at least one level higher score on the modified WHO ordinal scale.
  For SoC arm, no data were collected. Hence, 0 participants were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 1 | 0
Participants
  Baseline : WHO 7-point ordinal scale: 1 | 0 | 0
  Baseline : WHO 7-point ordinal scale: 2 | 0 | 0
  Baseline : WHO 7-point ordinal scale: 3 | 0 | 0
  Baseline : WHO 7-point ordinal scale: 4 | 1 | 0
  Baseline : WHO 7-point ordinal scale: 5 | 0 | 0
  Baseline : WHO 7-point ordinal scale: 6 | 0 | 0
  Baseline : WHO 7-point ordinal scale: 7 | 0 | 0
  Day 2 : WHO 7-point ordinal scale: 1 | 0 | 0
  Day 2 : WHO 7-point ordinal scale: 2 | 0 | 0
  Day 2 : WHO 7-point ordinal scale: 3 | 0 | 0
  Day 2 : WHO 7-point ordinal scale: 4 | 1 | 0
  Day 2 : WHO 7-point ordinal scale: 5 | 0 | 0
  Day 2 : WHO 7-point ordinal scale: 6 | 0 | 0
  Day 2 : WHO 7-point ordinal scale: 7 | 0 | 0
  Day 3 : WHO 7-point ordinal scale: 1 | 0 | 0
  Day 3 : WHO 7-point ordinal scale: 2 | 0 | 0
  Day 3 : WHO 7-point ordinal scale: 3 | 0 | 0
  Day 3 : WHO 7-point ordinal scale: 4 | 0 | 0
  Day 3 : WHO 7-point ordinal scale: 5 | 1 | 0
  Day 3 : WHO 7-point ordinal scale: 6 | 0 | 0
  Day 3 : WHO 7-point ordinal scale: 7 | 0 | 0

2. Secondary Outcome: Change in Room Air Oxygen Saturation (SpO2) From Baseline Over Time
Description: Pulse oximetry measurements were performed to evaluate SpO2. The effect of RESP301 as measured by room air SpO2 was assessed.
Time Frame: Day 1 (Baseline) Post-Nebulization, Day 2, 3, 4, 5, 6, and 7
Population: The intent-to-treat (ITT) population included all randomized participants. Here, the number analyzed in each row signified only the participants that were analyzed for each timepoint.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 11 | 5
Percent change
  Day 1 - Change from baseline | 0.1 (2.84) | NA (NA) — Post-dose nebulization did not occur in the SOC arm at Day 1. Soc arm data is not applicable.
  Day 2 - Change from baseline: number analyzed (Participants) | 9 | 2
  Day 2 - Change from baseline | -1.7 (4.09) | 1.5 (2.12)
  Day 3 - Change from baseline: number analyzed (Participants) | 8 | 3
  Day 3 - Change from baseline | 0.9 (2.80) | 3.3 (2.08)
  Day 4 - Change from baseline: number analyzed (Participants) | 5 | 3
  Day 4 - Change from baseline | 1.4 (2.61) | 3.0 (2.00)
  Day 5 - Change from baseline: number analyzed (Participants) | 4 | 3
  Day 5 - Change from baseline | 0.3 (1.26) | 4.0 (1.0)
  Day 6 - Change from baseline: number analyzed (Participants) | 2 | 2
  Day 6 - Change from baseline | -1.0 (1.41) | 4.5 (3.54)
  Day 7 - Change from baseline: number analyzed (Participants) | 2 | 0
  Day 7 - Change from baseline | 3.0 (2.83) |

3. Secondary Outcome: Change in National Early Warning Score (NEWS) 2 Symptom Score From Baseline Over Time
Description: The NEWS is based on a simple aggregate scoring system in which a score is allocated to physiological measurements, already recorded in routine practice, when patients present to, or are being monitored in hospital. Six simple physiological parameters form the basis of the scoring system: 1. Respiration rate; 2. Oxygen saturation; 3. Systolic blood pressure; 4. Pulse rate; 5. Level of consciousness or new confusion; 6. Temperature.
  Each score is 0-3 and individual scores are added together for an overall score. An additional two points are added if the patient is receiving oxygen therapy. The total possible score ranges from 0 to 20. The higher the score the greater the clinical risk. Higher scores indicate the need for escalation, medical review and possible clinical intervention, and more intensive monitoring.
Time Frame: Day 1 (Baseline), Day 2, 3, 4, 5, 6, and 7
Population: The intent-to-treat (ITT) population included all randomized participants. Here, the number analyzed in each row signifies only the participants who were analyzed for each time point.
Measure: Mean (Standard Deviation); unit: Score on a NEWS scale
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 12 | 5
Score on a NEWS scale
  Change from Baseline: Day 2 | -0.8 (1.99) | 1.4 (0.89)
  Change from Baseline: Day 3: number analyzed (Participants) | 9 | 5
  Change from Baseline: Day 3 | -1.3 (1.87) | -0.2 (1.3)
  Change from Baseline: Day 4: number analyzed (Participants) | 5 | 4
  Change from Baseline: Day 4 | 1.0 (2.55) | 0.5 (0.58)
  Change from Baseline: Day 5: number analyzed (Participants) | 4 | 4
  Change from Baseline: Day 5 | -2.0 (3.37) | -0.5 (3.11)
  Change from Baseline: Day 6: number analyzed (Participants) | 2 | 3
  Change from Baseline: Day 6 | -1.5 (2.12) | -2.0 (0.00)
  Change from Baseline: Day 7: number analyzed (Participants) | 2 | 0
  Change from Baseline: Day 7 | -1.0 (2.83) |

4. Secondary Outcome: Change From Baseline for Number of Participants on the Modified WHO Ordinal Scale at Each Visit
Description: A modified WHO ordinal scale was used for consistency with the recent study in adults hospitalized with severe COVID-19, to record the participant's status at the time of assessment. The modified WHO ordinal scale included the following levels :
  1= Not hospitalized, no limitations on activities; 2= Not hospitalized, limitation on activities; 3= Hospitalized, not requiring supplemental oxygen; 4= Hospitalized, requiring supplemental oxygen; 5= Hospitalized, on non-invasive ventilation or high-flow oxygen devices; 6= Hospitalized, on invasive mechanical ventilation or extra corporeal membrane oxygenation (ECMO); 7= Death. Higher scores mean worse outcome. Change from baseline for Number of Participants on the modified WHO ordinal scale was assesed.
Time Frame: Day 1 (Baseline), Day 2, 3, 4, 5, 6, and 7
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 12 | 5
Participants
  Day 2: change from baseline: Modified WHO 7-point ordinal scale -3 | 0 | 0
  Day 2: change from baseline: Modified WHO 7-point ordinal scale -2 | 0 | 0
  Day 2: change from baseline: Modified WHO 7-point ordinal scale -1 | 4 | 0
  Day 2: change from baseline: Modified WHO 7-point ordinal scale 0 | 8 | 5
  Day 2: change from baseline: Modified WHO 7-point ordinal scale 1 | 0 | 0
  Day 2: change from baseline: Modified WHO 7-point ordinal scale 2 | 0 | 0
  Day 2: change from baseline: Modified WHO 7-point ordinal scale 3 | 0 | 0
  Day 2: change from baseline: Modified WHO 7-point ordinal scale 4 | 0 | 0
  Day 3: change from baseline: Modified WHO 7-point ordinal scale -3: number analyzed (Participants) | 9 | 5
  Day 3: change from baseline: Modified WHO 7-point ordinal scale -3 | 0 | 0
  Day 3: change from baseline: Modified WHO 7-point ordinal scale -2: number analyzed (Participants) | 9 | 5
  Day 3: change from baseline: Modified WHO 7-point ordinal scale -2 | 3 | 1
  Day 3: change from baseline: Modified WHO 7-point ordinal scale -1: number analyzed (Participants) | 9 | 5
  Day 3: change from baseline: Modified WHO 7-point ordinal scale -1 | 1 | 0
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 0: number analyzed (Participants) | 9 | 5
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 0 | 4 | 4
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 1: number analyzed (Participants) | 9 | 5
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 1 | 1 | 0
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 2: number analyzed (Participants) | 9 | 5
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 2 | 0 | 0
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 3: number analyzed (Participants) | 9 | 5
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 3 | 0 | 0
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 4: number analyzed (Participants) | 9 | 5
  Day 3: change from baseline: Modified WHO 7-point ordinal scale 4 | 0 | 0
  Day 4: change from baseline: Modified WHO 7-point ordinal scale -3: number analyzed (Participants) | 5 | 4
  Day 4: change from baseline: Modified WHO 7-point ordinal scale -3 | 0 | 0
  Day 4: change from baseline: Modified WHO 7-point ordinal scale -2: number analyzed (Participants) | 5 | 4
  Day 4: change from baseline: Modified WHO 7-point ordinal scale -2 | 1 | 0
  Day 4: change from baseline: Modified WHO 7-point ordinal scale -1: number analyzed (Participants) | 5 | 4
  Day 4: change from baseline: Modified WHO 7-point ordinal scale -1 | 0 | 0
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 0: number analyzed (Participants) | 5 | 4
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 0 | 4 | 4
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 1: number analyzed (Participants) | 5 | 4
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 1 | 0 | 0
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 2: number analyzed (Participants) | 5 | 4
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 2 | 0 | 0
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 3: number analyzed (Participants) | 5 | 4
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 3 | 0 | 0
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 4: number analyzed (Participants) | 5 | 4
  Day 4: change from baseline: Modified WHO 7-point ordinal scale 4 | 0 | 0
  Day 5: change from baseline: Modified WHO 7-point ordinal scale -3: number analyzed (Participants) | 4 | 4
  Day 5: change from baseline: Modified WHO 7-point ordinal scale -3 | 0 | 0
  Day 5: change from baseline: Modified WHO 7-point ordinal scale -2: number analyzed (Participants) | 4 | 4
  Day 5: change from baseline: Modified WHO 7-point ordinal scale -2 | 2 | 1
  Day 5: change from baseline: Modified WHO 7-point ordinal scale -1: number analyzed (Participants) | 4 | 4
  Day 5: change from baseline: Modified WHO 7-point ordinal scale -1 | 0 | 2
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 0: number analyzed (Participants) | 4 | 4
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 0 | 2 | 1
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 1: number analyzed (Participants) | 4 | 4
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 1 | 0 | 0
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 2: number analyzed (Participants) | 4 | 4
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 2 | 0 | 0
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 3: number analyzed (Participants) | 4 | 4
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 3 | 0 | 0
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 4: number analyzed (Participants) | 4 | 4
  Day 5: change from baseline: Modified WHO 7-point ordinal scale 4 | 0 | 0
  Day 6: change from baseline: Modified WHO 7-point ordinal scale -3: number analyzed (Participants) | 2 | 2
  Day 6: change from baseline: Modified WHO 7-point ordinal scale -3 | 0 | 0
  Day 6: change from baseline: Modified WHO 7-point ordinal scale -2: number analyzed (Participants) | 2 | 2
  Day 6: change from baseline: Modified WHO 7-point ordinal scale -2 | 0 | 2
  Day 6: change from baseline: Modified WHO 7-point ordinal scale -1: number analyzed (Participants) | 2 | 2
  Day 6: change from baseline: Modified WHO 7-point ordinal scale -1 | 1 | 0
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 0: number analyzed (Participants) | 2 | 2
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 0 | 1 | 0
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 1: number analyzed (Participants) | 2 | 2
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 1 | 0 | 0
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 2: number analyzed (Participants) | 2 | 2
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 2 | 0 | 0
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 3: number analyzed (Participants) | 2 | 2
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 3 | 0 | 0
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 4: number analyzed (Participants) | 2 | 2
  Day 6: change from baseline: Modified WHO 7-point ordinal scale 4 | 0 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale -3: number analyzed (Participants) | 1 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale -3 | 0 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale -2: number analyzed (Participants) | 1 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale -2 | 1 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale -1: number analyzed (Participants) | 1 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale -1 | 0 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 0: number analyzed (Participants) | 1 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 0 | 0 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 1: number analyzed (Participants) | 1 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 1 | 0 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 2: number analyzed (Participants) | 1 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 2 | 0 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 3: number analyzed (Participants) | 1 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 3 | 0 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 4: number analyzed (Participants) | 1 | 0
  Day 7: change from baseline: Modified WHO 7-point ordinal scale 4 | 0 | 0

5. Secondary Outcome: Time to Improvement of at Least One Level Lower on the Modified WHO Ordinal Scale
Description: Time to improvement is the time in which the participant sees a decrease after first study treatment in the WHO 7-point ordinal scale from baseline to a value at least one level lower in days (date of decrease in WHO scale - first dose date + 1). In the case that a patient has not decreased in the WHO scale at time of analysis or withdraws from the study before leaving the hospital, they would be censored at their date of last assessment in the data cut or early discontinuation date, respectively.
Time Frame: From Baseline to Day 28
Population: The intent-to-treat (ITT) population included all randomized participants. Here, the Overall Number of Participants Analyzed signified only the participants who decrease by at least one level.
Measure: Median (Full Range); unit: Days
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 12 | 5
Days | 4.00 [2.00 to 10.50] | 5.00 [5.00 to 3.00]

6. Secondary Outcome: Time to Progression of at Least One Level Higher on the Modified WHO Ordinal Scale
Description: Time to progression is the time in which the patient sees an increase after first study treatment in the WHO 7-point ordinal scale from baseline to a value at least one level higher in days (date of increase in WHO scale - first dose date + 1). In the case that a patient has not increased in the WHO scale at time of analysis or withdraws from the study before leaving the hospital, they would be censored at their date of last assessment in the data cut or early discontinuation date, respectively.
Time Frame: From Baseline to Day 28
Population: The intent-to-treat (ITT) population included all randomized participants. Here, the Overall Number of Participants Analyzed signified only the participants who increase by at least one level.
Measure: Median (Full Range); unit: Days
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 1 | 0
Days | NA [NA to NA] — As only 1 participant was evaluable, hence Median and Full range is not calculable. |

7. Secondary Outcome: Number of Participants With Adverse Events
Description: AEs (non-serious) as variables of safety and tolerability of RESP301 were assessed.
  Severe AEs is defined as an event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event; and both AE and SAE can be assessed as severe.
Time Frame: From screening to safety follow up (Day 28)
Population: The safety analysis set includes the safety (SP) population would include all randomized participants who inhale any amount of study intervention or were randomized to the control arm. The SP would be analyzed according to the actual treatment received. This set will be used for the safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 14 | 5
Participants
  Participants with at least one AE | 10 | 2
  Participants with at least one AE of Grade 3 or higher | 1 | 0
  Participants with at least one treatment-related AE | 3 | 0
  Participants with at least one severe AE | 1 | 0
  Participants with at least one AE leading to study treatment withdrawal | 3 | 0
  Participants with at least one treatment-related AE leading to study treatment withdrawal | 1 | 0
  Participants with at least one AE leading to dose interruption | 1 | 0
  Participants with at least one treatment-related AE leading to dose interruption | 1 | 0

8. Secondary Outcome: Time to Hospital Discharge
Description: Time to hospital discharge is the time in the hospital after first study treatment in days (date of discharge - first dose date + 1). Patients who die before leaving the hospital would be considered failures (did not achieve hospital discharge) and censored. In the case that a patient is still hospitalized at time of analysis or withdraws from the study before leaving the hospital, they would be censored at their date of last assessment in the data cut or early discontinuation date, respectively.
Time Frame: Day 10
Population: The intent-to-treat (ITT) population included all randomized participants. Here, the Overall Number of Participants Analyzed signified only the participants who were discharged from hospital.
Measure: Median (Full Range); unit: Days
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 13 | 5
Days | 4.00 [3.00 to 6.00] | 6.00 [5.00 to 6.00]

9. Secondary Outcome: Number of Participants With Mortality by Day 28
Description: Incidence of mortality by Day 28 is the number of participants who have died by Day 28 and the percentage of patients reaching this endpoint will be summarized by treatment group.
Time Frame: Day 28
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 14 | 5
Participants | 0 | 0

10. Secondary Outcome: Reduction in Oxygen Saturation (SpO2) to <90%
Description: Room Air SpO2 for a summary of participants with reduction to < 90%, unless well clinically tolerated according to Investigator's opinion was assesed.
Time Frame: Day 1 (Baseline), Day 2, Day 3
Population: The intent-to-treat (ITT) population included all randomized participants. Here, the number analyzed in each row signified only the participants that were analyzed for each time point.
  Standard of Care (SoC) participants did not receive any nebulization. Hence, no participants were analyzed for Pre-nebulization and Post-nebulization. Therefore, no data were available.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 2 | 0
Percent change
  Day 1 Pre-Nebulization: number analyzed (Participants) | 1 | 0
  Day 1 Pre-Nebulization | 95.0 (NA) — As only 1 participant was evaluable, hence SD is not calculable. |
  Day 1 Post-Nebulization | 93.5 (2.12) |
  Day 2 Pre-Nebulization: number analyzed (Participants) | 1 | 0
  Day 2 Pre-Nebulization | 94.0 (NA) — As only 1 participant was evaluable, hence SD is not calculable. |
  Day 2 Post-Nebulization: number analyzed (Participants) | 1 | 0
  Day 2 Post-Nebulization | 86.0 (NA) — As only 1 participant was evaluable, hence SD is not calculable. |
  Day 3 Pre-Nebulization: number analyzed (Participants) | 1 | 0
  Day 3 Pre-Nebulization | 96.0 (NA) — As only 1 participant was evaluable, hence SD is not calculable. |
  Day 3 Post-Nebulization: number analyzed (Participants) | 1 | 0
  Day 3 Post-Nebulization | 94.0 (NA) — As only 1 participant was evaluable, hence SD is not calculable. |

11. Secondary Outcome: Events of Clinical Bronchial Hyper Responsiveness Related to Nebulization
Description: Incidence of clinical bronchial hyper responsiveness related to nebulization was assessed. Oxygen saturation decreased and wheezing was assessed as an incidence of clinical bronchial hyper-responsiveness related to nebulization, requiring temporal increase of supplemental oxygen.
Time Frame: From screening to safety follow up (Day 28)
Population: as for outcome 7
Measure: Number; unit: Events
Arm/Group | RESP301+SoC | Standard of Care (SoC)
Number analyzed (Participants) | 14 | 5
Events | 2 | 0

ADVERSE EVENTS:
Time Frame: From screening to safety follow up (30 days)
Description: Severe AEs is defined as an event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event; and both AE and SAE can be assessed as severe.
Groups:
- Standard of Care (SoC) Standard of Care (SoC): Participants received institutional SOC alone for the treatment of COVID-19.
Arm/Group | RESP301+SoC | Standard of Care (SoC) Standard of Care (SoC)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/5
Other Adverse Events (participants affected / at risk) | 10/14 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RESP301+SoC (N=14) | Standard of Care (SoC) Standard of Care (SoC) (N=5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Loss Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 2 (3) | 0 (0)
Liver Function Test Increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT04460183/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT04460183/SAP_001.pdf